CLINICAL TRIAL: NCT05585047
Title: Prospective Biomarkers for Treatment Response in Major Depressive Disorder
Brief Title: Treatment Response Biomarkers in MDD
Status: Recruiting | Type: Observational
Sponsor: Zhang Yan (Other)
Responsible Party: Sponsor-Investigator, Zhang Yan, Deputy Director of the National Clinical Research Center for Mental Disorders, Central South University
Organization: Central South University (Other)
Other Study IDs: MDD202011
Record Dates: First submitted 2022-10-15; First posted 2022-10-18 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Major Depressive Disorder
Keywords: Treatment Response; Biomarkers
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral venous blood，Faecal sample，hair
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This experiment intends to explore the differences among various types of depression, as well as the differences between healthy subjects and depressed patients, and find possible biological markers from the severity of symptoms, social function and cognitive function of depressed patients, combined with EEG characteristics, biological test indicators (blood, faeces, hair, etc.) and functional magnetic resonance imaging data.

To explore the changes in clinical symptoms, cognitive and social functions, and biological indicators of various types of patients before and after treatment, to provide references for the prognosis of various types, and to predict the future development of the disease according to the baseline indicators of patients; According to the above aspects, this experiment can follow up the patients with depression, track their disease development, and study the potential biological changes in the early stage of the disease, which has the potential to reveal the pathogenesis and provide guidance for the early diagnosis and intervention of depression.

DETAILED DESCRIPTION:
More specifically, the goals of this study are to 1) explore the potential biomarkers for Major Depressive Disorder by comparing MDD patients and healthy controls; 2) investigate the biochemical indicators for subtypes of MDD through long-term cohort follow-up studies; 3) investigate the differences and similarities among different types of MDD patients in terms of cognitive functions, biological tests, as well as neuroimaging data; 4) evaluate and analyze the prognosis of patients according to the baseline level, and search for the biomarkers regarding MDD treatment response to guide the clinical treatment and intervention of patients with MDD; 5) Through the long-term follow-up study, the behavioural and biochemical indicators of the patients with MDD were collected, the differences between the indicators before and after remission were examined, and the state and quality of the pathophysiological indicators of the patients with MDD were investigated.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is an outpatient/inpatient (but the subject who participated in the experimental treatment does not need to be hospitalized), and passed M.I.N.I. interview confirmed that the subjects met DSM-5 diagnostic criteria of current or past major depressive disorder.
2. Age 18-60 years old, regardless of gender;
3. Right-handed;
4. Junior high school education or above, capable of completing informed consent and cognitive test;
5. During the follow-up period, the subjects can take antidepressant treatment according to the doctor's advice of outpatient or resident.

   -

Exclusion Criteria:

1. Patients with psychotic symptoms;
2. M.I.N.I. was diagnosed as schizophrenia, schizophrenic affective disorder, schizophrenia-like disorder, Paranoia or current mental symptoms, post-traumatic stress disorder (currently or within the past year) or dysthymia;
3. with brain organic and serious physical diseases (such as thyroid disease, lupus erythematosus, diabetes, lung, liver and kidney) damage, infection, major trauma, etc.) exclude intracranial implants;
4. Clinically significant sensory disturbance that can't be corrected (for example, hearing impairment makes conversation impossible);
5. Pregnant and lactating women; -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Samples are taken from depressed patients in outpatient and inpatient departments of hospitals and recruited health care workers.
  480 subjects are expected to be collected and divided into two groups, 180 healthy subjects and 300 experimental subjects.
Sampling Method: Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Hamilton Depression Rating Scale-24 item (HAMD-24)Interview-based questionnaire used to measure the severity of depression | 8weeks
  Consists of 24 items with a score calculated. Higher scores are associated with more severe depression.

SECONDARY OUTCOMES:
Change in Hamilton Depression Rating Scale-17 item (HAMD-17)Interview-based questionnaire used to measure the severity of depression. | Baseline, 2weeks, 1 month, 2 months，4months，6months，1year
  Consists of 17 items with a score calculated. Higher scores are associated with more severe depression.
Change in Hamilton Anxiety Rating Scale-14 item (HAMA-14)Interview-based questionnaire used to measure the severity of anxiety. | Baseline, 2weeks, 1 month, 2 months，4months，6months，1year
  Consists of 14 items with a score calculated. Higher scores are associated with more severe anxiety.
Change in DSST (Number of Correct Symbols) | Baseline, 2weeks, 1 month, 2 months，4months，6months，1year
  Digit Symbol Substitution Test (DSST) is a cognitive test designed to assess psychomotor speed of performance requiring visual perception, spatial decision-making, and motor skills. It consists of 133 digits and requires the patient to substitute each digit with a simple symbol in a 90-second period. Each correct symbol is counted, and the total score ranges from 0 (less than normal functioning) to 133 (greater than normal functioning)." as a description of DSST.
Change in Generalized Anxiety Disorder-7 (GAD-7) | Baseline, 2weeks, 1 month, 2 months，4months，6months，1year
  The GAD-7 aims to assesses the severity of anxious symptoms.
Change in Patient Health Questionnaire-9 (PHQ-9) | Baseline, 2weeks, 1 month, 2 months，4months，6months，1year
  The PHQ-9 aims to assesses the severity of depression symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Central South University, Changsha, Hunan, China